CLINICAL TRIAL: NCT03896594
Title: A Dose Block-randomized, Double-blind, Placebo Controlled, Dose-escalation Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetics After Multiple Oral Dose of HL237 in Healthy Male Subject
Brief Title: A Multiple Dose of HL237 in Healthy Male Subject
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: HL237-102
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HL237 200mg (Experimental): HL237 100mg 1 tablet twice a day
  Interventions: Drug: HL237; Drug: Placebo Oral Tablet
- HL237 400mg (Experimental): HL237 100mg 2 tablets twice a day
  Interventions: Drug: HL237; Drug: Placebo Oral Tablet
- HL237 800mg (Experimental): HL237 400mg 1 tablet twice a day
  Interventions: Drug: HL237; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: HL237 — Experimental
Drug: Placebo Oral Tablet — placebo with same properties except for active ingredient

SUMMARY:
HL237 is a new autoimmune therapeutic agent for rheumatoid arthritis, including the basic structure of biguanide in metformin, an existing diabetes drug.

The immune modulating activity of HL237 was demonstrated in animal model. HL237 is a STAT3 inhibitor and STAT3 is well known for an important regulator inhibiting Th17 cells and activating Treg cells.

Therefore, when STAT3 activity is inhibited, it is expected to be able to treat autoimmune diseases such as rheumatoid arthritis.

This is the first repeated administration clinical trial performed for the development of HL237 and is intended to evaluate the safety, tolerability and pharmacokinetics of each dose group.

DETAILED DESCRIPTION:
Doses are increased sequentially from low-capacity groups, and within six weeks after the last dose of the last subject in the ongoing dose phase, if available pharmacokinetic data are judged acceptable under review by investigators, sponsor and safety review committees, then proceed to the next dose stage.

ELIGIBILITY:
Inclusion Criteria:

* A healthy adult male aged 20 years or older and 45 years old at the time of the screening test
* Those who weigh more than 55kg but weigh less than ± 20% of ideal body weight
* Proper contraception during the clinical trial period
* After hearing the detailed explanation of the clinical trial, those who decide to participate voluntarily and write agreement

Exclusion Criteria:

* Clinically significant, a person with a history of neurological, psychiatric, malignant, cardiovascular, respiratory, kidney, endocrine, hematologic, digestive or central disease
* a person with a history of gastrointestinal disorders that may affect the absorption of pharmaceuticals for clinical trials (Crohn's disease, ulcers, etc.) or gastrointestinal surgery (except for simple cecal surgery or hernia surgery)
* a person with a history of hypersensitivity or clinically significant hypersensitivity to the clinical trial drug or additives
* a person judged to be inappropriate for the subject by health screening (history of disease, physical examination, vital signs, electrocardiogram, laboratory test, etc.)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-12-24 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | 14days after administration
  maximum serum concentration after the drug has been administrated
Area Under the Curve [AUC] | 14days after administration
  AUC after the drug has been administrated
Half life [t1/2] | 14days after administration
  Half life after the drug has been administrated

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 14days after administration
  Adverse Adverse Events, Serious Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul, Seocho-gu, South Korea